CLINICAL TRIAL: NCT04382482
Title: Remotely Controlled Intervention for Developmental Reading and Spelling Disorders
Brief Title: Remotely Controlled Intervention for Developmental Reading and Spelling Disorders Through the Tachidino Platform
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: 08/17oss
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Developmental Dyslexia; Developmental Spelling Disorder
Keywords: Developmental Dyslexia; Intervention; Hemisphere-specific stimulation; Visual-attentional training; E-health; telerehabilitation; web-based platform; Developmental Spelling Disorder
MeSH Terms: conditions — Dyslexia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tachidino: This group is being treated through the web platform Tachidino for remote rehabilitation of reading and spelling disorders
  Interventions: Device: Tachidino

INTERVENTIONS:
Device: Tachidino — Web-platform delivering remote treatment of reading and spelling disorders through the (visual or auditory) presentation of words and sentences to be either decoded or corrected (reordering wrong letter sequences).

SUMMARY:
The study aims to document the effects of the intervention system for specific reading and spelling disorders, currently in use at Scientific Institute (IRCCS) Medea as an innovative intervention model in e-health mode. The model constitutes the application of research data collected in more than fifteen years research on the causes of dyslexia and rehabilitation techniques, combined with the most advanced technologies for remotely-controlled clinical management and therapy monitoring through adaptive, self-updating algorithms.

A single group of about 80 children will be observed and their performance on reading, spelling and metaphonological tests at pre-test, post-test and follow-up (after 6 months) will be recorded in order to assess improvement (and, consequently, treatment effectiveness) and its stability. The improvements obtained in four weeks treatment will subsequently be compared with those obtained with outpatient intervention programmes of the same duration and intensity.

DETAILED DESCRIPTION:
The system for the improvement of reading and writing skills ("Tachidino" software) is based on two principles of proven effectiveness:

1. The selective stimulation of a cerebral hemisphere and specific reading strategies. Taking up some of the principles already set out in the Balance Model of Dyslexia, the aim is to retrace the different stages of reading acquisition by focusing on those stages and processes which have proved more problematic or less efficiently activated. Such stages may require greater involvement of the right hemisphere, carrying out an accurate visual analysis of the material to be read, or of the left hemisphere, anticipating the words to be read by exploiting linguistic skills (knowledge of words, relationships between meanings, relationships between sounds, grammatical agreement and syntactic rules, etc.);
2. the training of selective visuospatial attention, as well as the perception of rapid movement and the analysis of the visual characteristics of words. A further mechanism involved in the training is the so-called visual crowding, an automatic effect of our perceptual system producing a sort of "blurring" of the visual areas surrounding the object to be analyzed, to make its vision clearer. A malfunction of this mechanism and an insufficient ability to concentrate visual attention in a restricted area of the visual field, or to move it quickly and precisely from one point to another would be among the causes of reading disorders, as suggested by the Magnocellular theory of dyslexia.

Studies carried out by researchers at IRCCS Medea have shown excellent results for the two types of treatment (Hemisphere-specific stimulation according to the Balance Model, and Visual-attentional training with Action Video- Games or Wii games, but above all they showed how these effects are strongly enhanced by the association in a single intervention.

Clinical and assessment procedures

In the Tachidino program, the child (sitting in fron of the computer screen) is required to recognize the target candy (a spiral candy) among various candies (distractors) and press the space bar at the exact moment the target candy is crossing a circle target (fixation point). The word to be decoded/encoded is presented, visually or auditory, only if the child clicks at the right moment, thus ensuring that fixation was in correspondence with the fixation point in the center of the visual field. If the bar is pressed in the target timeframe and in correspondence of the target candy, the word to be decoded/encoded is immediately presented and the child is asked to either write the word on the keyboard or re-order a sequence containing all the correct graphemes in random order.

All visual stimuli are presented at tachistoscopic speed to a visual hemifield in order to stimulate the contralateral hemisphere to a greater degree, or they may also be flashed in the center of the computer screen, involving both hemispheres simultaneously.

The visual hemisphere-specific stimulation is based on a revisit of Bakker's 'Balance model'. Each child was classified as a P-, L-, or M-type dyslexic reader based on the persistent over-reliance on specific reading strategies as shown by reading and spelling errors, and on reading speed.

As per current clinical practice, intervention in "e-health" mode is divided into one or more rehabilitation modules through the use of the Tachidino platform, with systematic monitoring and motivational reinforcement by professionals with experience in e-health approaches. In order to be included in the training, the child must have already obtained a diagnosis of dyslexia, according to the current diagnostic standards.

The structure of the intervention modules, as currently implemented, is as follows:

* 1 initial meeting to get to know the child, pre-test assessment - reading and writing tests of words, non-words and sentences, metaphonological tests (phonemic elision and synthesis) and text reading tests (reading accuracy and speed) in order to define dyslexia subtypes; intervention planning - demonstration of Tachidino use and programming of first activities
* telephone support to monitor and motivate correct use of the software, during active intervention
* 1 final assessment meeting (with repetition of the tests used at pre-test and compilation of satisfaction questionnaires).
* 1 follow-up meeting 6 months after discharge with repetition of reading tests (this meeting is relevant in order to assess stabilization of obtained improvements)

Participants' characteristics: Children aged between 7 and 14 years with a diagnosis of Specific Reading Disorder or Specific Spelling Disorder, not treated before.

The improvements obtained in one month treatment will be compared with those obtained with outpatient intervention programmes of the same duration and intensity, combining treatment based on the two component parts: Visual Hemisphere-Specific Stimulation (V-HSS) and Visual-Attentional Training with Action Video Games.

ELIGIBILITY:
Inclusion Criteria:

* A formal diagnosis of Developmental Dyslexia, Specific Reading Disorders, Specific Spelling Disorders or Mixed Learning Disorders
* Age between 7 and 16
* Attending at least the third class of primary school
* Monolingual speakers of Italian or bilingual speakers with perfect mastery of the Italian language (equivalent to monolinguals)
* Intelligence Quotient (IQ) >= 80
* At least one z-score below -2 Standard Deviations from age mean in at least one of the following tests: text reading, word reading, nonword reading, word writing to dictation, nonword writing to dictation ("DDE-2" battery, "MT" tests)
* Not having received any specific rehabilitation treatment for dyslexia before

Exclusion Criteria:

* Intellectual disability
* Neurological disorders
* Sensory deficits that are not /cannot be corrected-to-normal by lenses or hearing aids.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited among those referred to IRCCS Medea because of learning and school-achievement problems. All children who were offered treatment through the web-based platform "Tachidino" and who met inclusion/exclusion criteria were enrolled in the study after their parents had accepted and signed informed consent.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
change from pre-test to post-test in reading ability | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in reading measures (speed and accuracy in word, nonword and text reading standardized tests: Memory Training (MT) group reading test and "Developmental Dyslexia and Dysgraphia (DDE-2); average of the scores expressed as z-scores with respect to age norms)
change from pre-test to post-test in spelling ability | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in spelling tests (writing to dictation of words, nonwords and sentences) - average of the scores expressed as z-scores with respect to age norms in standardized tests ("DDE-2", "Diagnosis of Dysgraphic Disorders" (DDO-2))

SECONDARY OUTCOMES:
change from pre-test to post-test in metaphonological ability | 4 weeks
  Difference in treatment-related changes (post-test minus pre-test) observed in metaphonological tests (phonemic elision and phoneme blending) - average of the number of errors in the two tests
persistence of improvement at follow-up (6 months) | 7 months (1 month intervention and 6 months follow-up)
  no significant difference between post-test scores and follow-up scores (follow-up 6 months after discharge and in the absence of further intervention) in text, word and nonword reading ("MT" tests, "DDE-2")
satisfaction with remote intervention experience | 4 weeks
  scores expressed by parents and patients at post-test, on a questionnaire concerning satisfaction with the delivery of remote intervention and its effects

OTHER OUTCOMES:
comparison with existing data about inpatient treatment effectiveness | 4 weeks
  difference in z-scores (reading speed and accuracy measured with "MT tests" and "DDE-2") between changes obtained with Tachidino remotely delivered intervention and inpatient treatment with the same combined components (Visual Hemisphere-Specific Stimulation and Action Video-Games), both conducted over 4 weeks. Data about improvement obtained with inpatient treatment were previously collected at IRCCS E. Medea (ClinicalTrials.gov NCT02791841, published in Frontiers in Psychology, 2020)

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Lorusso, Ph.D., Principal Investigator — IRCCS E. Medea
Locations (1):
- Scientific Institute IRCCS E. Medea, Bosisio Parini, LC, Italy

REFERENCES:
- [Background] Bakker DJ. Neuropsychological classification and treatment of dyslexia. J Learn Disabil. 1992 Feb;25(2):102-9. doi: 10.1177/002221949202500203. PMID 1583415
- [Background] Bakker DJ. Treatment of developmental dyslexia: a review. Pediatr Rehabil. 2006 Jan-Mar;9(1):3-13. doi: 10.1080/13638490500065392. PMID 16352500
- [Background] Lorusso ML, Facoetti A, Paganoni P, Pezzani M, Molteni M. Effects of visual hemisphere-specific stimulation versus reading-focused training in dyslexic children. Neuropsychol Rehabil. 2006 Apr;16(2):194-212. doi: 10.1080/09602010500145620. PMID 16565034
- [Background] Franceschini S, Gori S, Ruffino M, Viola S, Molteni M, Facoetti A. Action video games make dyslexic children read better. Curr Biol. 2013 Mar 18;23(6):462-6. doi: 10.1016/j.cub.2013.01.044. Epub 2013 Feb 28. PMID 23453956
- [Background] Lorusso ML, Facoetti A, Bakker DJ. Neuropsychological treatment of dyslexia: does type of treatment matter? J Learn Disabil. 2011 Mar-Apr;44(2):136-49. doi: 10.1177/0022219410391186. PMID 21383106
- [Result] Lorusso ML, Borasio F, Molteni M. Remote Neuropsychological Intervention for Developmental Dyslexia with the Tachidino Platform: No Reduction in Effectiveness for Older Nor for More Severely Impaired Children. Children (Basel). 2022 Jan 5;9(1):71. doi: 10.3390/children9010071. PMID 35053699
- [Result] Lorusso ML, Borasio F, Misto P, Salandi A, Travellini S, Lotito M, Molteni M. Remote treatment of developmental dyslexia: how ADHD comorbidity, clinical history and treatment repetition may affect its efficacy. Front Public Health. 2024 Jan 10;11:1135465. doi: 10.3389/fpubh.2023.1135465. eCollection 2023. PMID 38269376
- [Result] Lorusso ML, Borasio F, Molteni M. The challenge of remote treatment in neuropsychological intervention for reading and spelling in dyslexia: A prospective observational cohort study. Dyslexia. 2024 Feb;30(1):e1758. doi: 10.1002/dys.1758. Epub 2024 Jan 15. PMID 38224428